CLINICAL TRIAL: NCT01766245
Title: A Randomised, Single Centre, Double-blind, Two-period, Cross-over Trial in Healthy Subjects Investigating the Bioequivalence Between Subcutaneous Injections of Semaglutide Produced by Two Manufacturing Processes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-4010; 2012-002212-20 (EudraCT Number); U1111-1130-3931 (Other: WHO)
Record Dates: First submitted 2012-12-19; First posted 2013-01-11 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes; Healthy
Keywords: mm
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation A followed by Formulation B (Experimental)
  Interventions: Drug: semaglutide
- Formulation B followed by Formulation A (Active Comparator)
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — For subcutaneous (s.c., under the skin), single dose administration at two separate dosing visits.

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the bioequivalence (assessment of the expected biological equivalence of two pharmaceutical drug products with identical active ingredient) between subcutaneous injections of semaglutide produced by two manufacturing processes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Body mass index (BMI) of 18.5-30 kg/m^2 (both incl.)

Exclusion Criteria:

* History of or presence of cancer, diabetes, pancreatitis or any clinically relevant cardiovascular diseases or other major disorders
* Use of prescription or non-prescription medicinal products (except routine vitamins, acetylsalicylic acid and paracetamol) within 3 weeks (or within 5 half-lives of the medicinal product, whichever is longest) prior to the first dosing of semaglutide
* Smoking, drug or alcohol abuse
* Female of childbearing potential who is pregnant, breast-feeding or intend to become pregnant or not using adequate contraceptive methods for the duration of the trial and for 3 months following the last dose of semaglutide

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma semaglutide concentration curve | 0-4 weeks after a single dose s.c. semaglutide administration
Cmax, the maximum plasma semaglutide concentration | 20-40 hours after a single dose s.c. semaglutide administration

SECONDARY OUTCOMES:
The area under the plasma semaglutide concentration curve | From time 0 to infinity after a single dose s.c. semaglutide administration
tmax, time to Cmax of semaglutide | 20-40 hours
t½, terminal elimination half-life of semaglutide | 140-200 hours
Incidence of adverse events (AEs) | From first dosing to follow-up (5-7 weeks after the second dosing)
Hypoglycaemic episodes | From first dosing to follow-up (5-7 weeks after the second dosing)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Berlin, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com